CLINICAL TRIAL: NCT05684887
Title: Digital Tools to Expand COVID-19 Testing in Exposed Individuals in Cameroon (DTECT Cameroon)
Brief Title: Digital Tools to Expand COVID-19 Testing in Exposed Individuals in Cameroon
Acronym: DTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Find (Other); Cameroon Ministry of Public Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EG0284
Record Dates: First submitted 2023-01-09; First posted 2023-01-13 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: COVID-19; Contact Tracing; mHealth
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized trial conducted in eight (8) Health Districts with a high number of people being tested for SARS-CoV-2 in the Littoral region in Cameroon, comparing two strategies for COVID-19 contact tracing of SARS-CoV-2 infected index patients:
  * The standard of care (SOC) implements the contact tracing using a manual process based on current routine approach (use of the Mamal Pro application without digital contact tracing module).
  * The intervention (ITV) will implement the contact tracing using a digitalized process (addition of the Mamal Pro digital contact tracing module to the Mamal Pro app).
  The randomization unit (cluster) will be the district with selected testing units and/or health facilities where SARS-CoV-2 infected patients (index cases) are diagnosed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care model (SOC) (No Intervention): This model is based on the standard of care recommended by the Cameroon National COVID-19 response program.
- Intervention model (ITV) (Experimental): Implementation of the contact tracing using a digitalized process (addition of the Mamal Pro digital contact tracing module to the Mamal Pro app).
  Interventions: Other: Digital based contact tracing

INTERVENTIONS:
Other: Digital based contact tracing — * Listing of contacts by SARS-CoV-2 positive individuals in Mamal Pro app + verification and validation by a health care worker.
  * Immediate access to the contact list in Mamal Pro once validated by the health care worker.
  * Contacts are immediately notified by text message automatically sent to all contacts with phone numbers and later called by the HCWs responsible for carrying out the contact tracing at the district level.
  * Contacts will be invited to go to the nearest testing facilities/units to get tested.
  * Those who are unable or refuse to come for testing are followed up by phone for 10 days for the occurrence of COVID-19 symptoms.
  * Information about the contact tracing process during communication with contacts are recorded in Mamal Pro digital contact tracing module.
  Arms: Intervention model (ITV)

SUMMARY:
According to the WHO, contact tracing - along with robust testing, isolation, and care of cases is a key strategy for interrupting chains of transmission of SARS-CoV-2 and reducing mortality associated with COVID-19. Contact tracing, however, has a number of challenges. These include incomplete identification of contacts, inefficiencies in paper-based reporting systems, complex data management requirements, and delays in the identification of contacts and testing of contacts. In many settings, contact tracing has proven to be too resource-intensive to implement at scale, especially with higher levels of community transmission, highlighting the need for more efficient contact tracing approaches. Digital tools afford the possibility of strengthening contact tracing for COVID-19, in a more efficient way. However, there is limited evidence of the effectiveness and impact of these tools in the COVID-19 response, including contact tracing.

This study proposes to compare the cascade of care between two strategies for COVID-19 contact tracing of SARS-CoV-2 infected index patients in Cameroon. In one strategy (intervention), the health facilities and health district testing units will implement contact tracing using a digital tool developed to support the tracing and testing of contacts (addition of a digital contact tracing module to the main platform for COVID-19 testing in Cameroon (Mamal Pro app)). This strategy will be compared to the standard contact tracing process (control), based on the current routine approach (use of the Mamal Pro application without the digital contact tracing module).

DETAILED DESCRIPTION:
The study's general objective is to assess the effectiveness, feasibility, acceptability, and cost associated with the addition of a Mamal Pro digital contact tracing module to the Mamal Pro app in improving COVID-19 contact tracing and testing in Littoral, Cameroon.

Specific objectives are:

1. Primary objective: To determine the effectiveness of the use of a Mamal Pro digital contact tracing module added to the Mamal Pro app in improving COVID-19 contact tracing and testing compared to the SOC as measured by:

   * The number and proportion of reported contacts who received SARS-CoV-2 testing.
   * The number and proportion of contacts who are successfully reached by phone by MOH district contact tracing unit.
   * The number and proportion of contacts testing positive for SARS-CoV-2 infection.
   * The time from SARS-CoV-2 infected index patient identification of contacts to communication with the contact by the district contact tracing unit.
2. Secondary objectives:

   * To assess the feasibility and acceptability of the use of the Mamal Pro digital contact tracing module through structured interviews with MOH facility staff, district unit contract tracing teams, and individuals undergoing SARS-CoV-2 testing.
   * To estimate the total cost of using the Mamal Pro contact tracing module for tracing SARS-CoV2 positive case contacts and cost per contact traced using the module.

ELIGIBILITY:
Inclusion Criteria:

* All contacts listed by individuals registered in the Mamal Pro app for testing, who test positive for SARS-CoV-2 in the selected health district testing units and health facilities in Cameroon.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Successful contact tracing | 10 days
  The primary outcome is the proportion of contacts declared by the index case who are successfully called by the district contact tracing unit and the proportion of contacts who receive SARS-CoV-2 testing, as per MOH standard testing procedures.

SECONDARY OUTCOMES:
Contacts testing positive for SARS-CoV-2 infection. | 10 days
  The proportion of contacts testing positive for SARS-CoV2 infection
Feasibility of the intervention model of contact tracing | 4 months
  * ease of use
  * time to complete the process in the Mamal Pro digital contact tracing module
  * integration with other clinic activities
Acceptability intervention model of contact tracing by the index cases (negative and positive) and health care workers | 4 months
  * satisfaction of using the Mamal Pro digital contact tracing module compared with the usual standard of care approach
  * challenges with this approach to contact tracing
  * suggestions for improvement.
Cost of the intervention | 4 months
  Cost estimates for using Mamal Pro digital contact tracing module to trace contacts, and cost per contact traced.
Timely communication with contacts | 4 months
  Time (days) between receipt of contact list and contacts' call attempts
SMS sent | 4 months
  Proportion of SMS delivered, (numerator: SMS sent, denominator: phone numbers)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Tchakounte Youngui, MD, MPH, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation; Godfrey Woelk, PhD, MCOMMH, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (22):
- Cameroon (22):
  - Bonanjo Integrated Health Center, Douala, Littoral Region
  - Bonassama District COVID testing unit, Douala, Littoral Region
  - Bonassama district hospital, Douala, Littoral Region
  - Cité des palmiers District COVID testing unit, Douala, Littoral Region
  - Cité des palmiers district hospital, Douala, Littoral Region
  - CMA Bonamoussadi, Douala, Littoral Region
  - CMA Nyala, Douala, Littoral Region
  - CMA Soboum hospital, Douala, Littoral Region
  - Deido District COVID testing unit, Douala, Littoral Region
  - Deido district hospital, Douala, Littoral Region
  - General Hospital Douala, Douala, Littoral Region
  - Gynecological-Obstetric and Pediatric Hospital Douala (HGOPED), Douala, Littoral Region
  - Japoma District COVID testing unit, Douala, Littoral Region
  - Laquintinie Hospital, Douala, Littoral Region
  - Logbaba District COVID testing unit, Douala, Littoral Region
  - Logbaba district hospital, Douala, Littoral Region
  - Mbangue District COVID testing unit, Douala, Littoral Region
  - Mboppi Baptist hospital, Douala, Littoral Region
  - New Bell District COVID testing unit, Douala, Littoral Region
  - New Bell district hospital, Douala, Littoral Region
  - Nylon District COVID testing unit, Douala, Littoral Region
  - Nylon district hospital, Douala, Littoral Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Songane M, Tchakounte Youngui B, Mambo A, Bonabe G, Djikeussi T, Epee E, Tsigaing PN, Ndongo MLA, Mayap Njoukam C, Kana R, Tenkeu SZ, Simo L, Kouatchouang AV, Machekano R, Zoung-Kanyi Bissek AC, Tchendjou P, Tiam A, Guay L, Suleiman K, Akinwusi O, Kadam R, Akugizibwe P, Mukherjee S, Woelk G, Tchounga B. Using an app for COVID-19 contact tracing costs less per person traced than manual tracing: microcosting analysis of a randomised trial in Cameroon. BMJ Public Health. 2025 Jan 21;2(Suppl 1):e001064. doi: 10.1136/bmjph-2024-001064. eCollection 2024 Jul. PMID 40017704
- [Derived] Tchakounte Youngui B, Mambo A, Machekano R, Kana R, Epee E, Tenkeu SZ, Tsigaing PN, Ndongo MLA, Njoukam CM, Bichara L, Katcho TD, Mbunka MA, Longla TA, Simo L, Kouatchouang AV, Tchendjou P, Tiam A, Guay L, Suleiman K, Akinwusi O, Kadam R, Akugizibwe P, Songane M, Woelk G, Tchounga BK; DTECT study group. Improving COVID-19 contact tracing and testing of exposed individuals in Cameroon using digital health technology: a cluster randomised trial. EClinicalMedicine. 2024 Jul 13;74:102730. doi: 10.1016/j.eclinm.2024.102730. eCollection 2024 Aug. PMID 39109192